CLINICAL TRIAL: NCT06548698
Title: The Impact of Escape Room Experience on Problem Solving and Professional Behavior Levels in Nursing Students: An Interventional Educational Study
Brief Title: The Impact of Escape Room Experience in Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Seda Akutay, Research Assistant, TC Erciyes University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ErciyesUniv
Record Dates: First submitted 2024-08-01; First posted 2024-08-12 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Nursing Education
Keywords: nursing students; nursing education; escape room; problem solving; professional behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Other: escape room
- Control group (No Intervention)

INTERVENTIONS:
Other: escape room — Nursing students in the intervention group analyzed the breast cancer surgery case with the escape room experience.
  Arms: Intervention group

SUMMARY:
Gamification is an applied, team-based approach in which students are actively involved. This study was conducted to evaluate the effect of escape room experience on the level of problem solving skills and professional behavior in nursing students.

This study was completed in a randomized controlled trial with 43 final year nursing students from a university. Students were randomized into intervention (n=22) and control (n=21) groups. In this study, data were collected with the Game Experience Scale, Problem Solving Inventory, and Nursing Students Professional Behavior Scale. The data obtained from the study were evaluated with SPSS 24.0. Descriptive statistics; number (n), percentage (%), mean (X), standard deviation (SD) were given. Statistical significance level was evaluated as p<0.05. The students in the intervention group analyzed the breast cancer surgery case with the escape room experience. The students were divided into groups of 5 and tried to complete the tasks given by the researchers within 30 minutes. During the escape room practice, the researchers were present in the rooms as observers and evaluated the participants.

ELIGIBILITY:
Inclusion Criteria:

* Active students in the spring semester of the 2023-2024 academic year,
* A fourth-year nursing student,
* To take the surgical diseases nursing intern practice module,
* Preparing an individualized patient care plan for at least one surgical patient,
* Students who have previously prepared and presented at least one surgical patient-specific case with group work

Exclusion Criteria:

* Those who have lessons they did not take in 1st-3rd classes,
* Never planned care for surgical patients in previous clinical practice,
* Students who refused to participate in the study

Ages: 21 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2024-05-06 (Actual); Primary Completion 2024-06-12 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Problem solving level | 5 week
  The problem solving levels of nursing students will be evaluated using the problem solving inventory in the first week and the last week of the 5-week follow-up period.
professional behavior level | 5 week
  The professional behavior levels of nursing students will be evaluated using the Professional Behavior Scale for Nursing Students in the first and last week of the 5-week follow-up period.

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University Faculty of Health Sciences, Kayseri, Kayseri, Turkey (Türkiye)